CLINICAL TRIAL: NCT03716466
Title: Evaluation of Prophylactic Endotracheal Intubation in the Patients With Upper Gastrointestinal Bleeding Undergoing Urgent Endoscopy: A Prospective Observational Study
Brief Title: Evaluation of Prophylactic Endotracheal Intubation
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Dawood Nasir, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU 072018-045
Record Dates: First submitted 2018-09-28; First posted 2018-10-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Intubation;Difficult; Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endotracheal intubation: Cases with prophylactic endotracheal intubation during urgent endoscopy procedure for upper gastrointestinal bleeding .
  Interventions: Other: Endotracheal intubation
- No airway intervention: Cases without airway intervention during urgent endoscopy procedure for upper gastrointestinal bleeding
  Interventions: Other: No airway intervention

INTERVENTIONS:
Other: Endotracheal intubation — Subjects will receive prophylactic endotracheal intubation for upper gastrointestinal endoscopy procedure
  Groups: Endotracheal intubation
Other: No airway intervention — Subjects without prophylactic endotracheal intubation during upper gastrointestinal endoscopy procedure
  Groups: No airway intervention

SUMMARY:
Upper gastrointestinal (GI) bleeding is defined as patients who either presented with hematemesis or presented with melena along with evidence of hemodynamic compromise. These patients have risk of aspiration of blood along with gastric content. The mortality rate can be 15% to 20% in the cases with variceal bleeding. From a practical standpoint, it is widely accepted that the best way to secure an airway during upper GI bleeding is prophylactic endotracheal intubation (PEI). The aim of this study is to determine the incidence of complications among critically ill patients with upper GI bleeding and received urgent endoscopy.

DETAILED DESCRIPTION:
This is a prospective observational study. After IRB approval, consecutive patient with upper GI bleeding and undergoing urgent endoscopy will be enrolled to the study over 24 months period. Data pull will be requested from Parkland Office of Research Administration (ORA) regarding eligible subjects and protocol requiring data elements. The data pull will be requested at the end of the 24 months-period.

Primary endpoint:

The incidence of cardiovascular unplanned event within 48 hours of the upper gastrointestinal endoscopy procedure.

Secondary end points:

The incidence of pulmonary unplanned event within 48 hours of the upper gastrointestinal endoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Presence of upper gastrointestinal bleeding either presented with hematemesis or melena along with evidence of hemodynamic compromise.
* Received procedural (conscious) sedation
* Undergoing urgent upper gastrointestinal endoscopy procedures

Exclusion Criteria:

* Intubation other than airway protection
* Prior tracheostomy before onset of gastrointestinal bleeding
* Subjects intubated before transfer to gastrointestinal suite
* Subjects without hemodynamic instability
* Subjects with a diagnosis of pneumonia, acute respiratory distress syndrome, myocardial infarction, pulmonary edema, arrhythmia, or cardiac arrest before endoscopy
* Endoscopy done for other than upper gastrointestinal bleeding
* Pregnant subjects

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cases with upper gastrointestinal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Cardiovascular unplanned event | Postoperative up to 48 hours
  The number of cardiovascular unplanned event after upper gastrointestinal endoscopy, up to 48 hours

SECONDARY OUTCOMES:
Pulmonary unplanned event | Postoperative up to 48 hours
  The number of pulmonary unplanned event after upper gastrointestinal endoscopy, up to 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: David Nasir, MD, Study Director — 214-590-5352
Locations (1):
- Parkland Health Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No